CLINICAL TRIAL: NCT06682793
Title: A Seamless Phase 1/2 Study to Evaluate the Safety and Efficacy of A2B395, an Allogeneic Logic-gated Tmod™ CAR T, in Heterozygous HLA-A*02 Adults With Recurrent Unresectable, Locally Advanced, or Metastatic Solid Tumors That Express EGFR and Have Lost HLA-A*02 Expression
Brief Title: A Study to Evaluate the Safety and Efficacy of A2B395, an Allogeneic Logic-gated CAR T, in Participants With Solid Tumors That Express EGFR and Have Lost HLA-A*02 Expression
Acronym: DENALI-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: A2 Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2B395-101
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor, Adult; Colorectal Cancer; Non-Small Cell Lung; NSCLC (Non-small Cell Lung Cancer); Cancer; Colon Cancer; Rectal Cancer; Lung Cancer; CRC; Head and Neck Squamous Cell Cancer; HNSCC; Renal Cell Carcinoma; RCC; Kidney Cancer; Triple Negative Breast Cancer; TNBC; Colorectal Adenocarcinoma
Keywords: CAR T Cell; Solid Tumors; Allogeneic; T Cell; EGFR; HLA-A2; Solid tumors expressing EGFR; CRC; Colorectal; Cell Therapy; Gene Therapy; Blocker; Cancer; NSCLC; Non small Cell Lung Cancer; Lung Cancer; renal cell carcinoma; RCC; Kidney Cancer; Renal cell cancer; Triple negative breast cancer; TNBC
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Lung Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Kidney Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- A2B395 (Experimental): Participants receive preconditioning lymphodepletion (PCLD) regimen followed by a single dose of A2B395 intravenously on day 0
  Interventions: Biological: A2B395; Diagnostic Test: xT CDx with HLA-LOH assay

INTERVENTIONS:
Biological: A2B395 — Allogeneic logic-gated Tmod CAR T cells
  Other Names: Tmod CAR T-cell Therapy
Diagnostic Test: xT CDx with HLA-LOH assay — An investigational next generation sequencing (NGS) in vitro diagnostic (IVD) medical device

SUMMARY:
The goal of this study is to test A2B395, an allogeneic logic-gated Tmod™ CAR T-cell product in subjects with solid tumors including colorectal cancer (CRC), non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), triple-negative breast cancer (TNBC), renal cell carcinoma (RCC) and other solid tumors that express EGFR and have lost HLA-A*02 expression.

The main questions this study aims to answer are:

* Phase 1: What is the recommended dose of A2B395 that is safe for patients
* Phase 2: Does the recommended dose of A2B395 kill the solid tumor cells and protect the patient's healthy cells

Participants will be required to perform study procedures and assessments, and will also receive the following study treatments:

* Enrollment in BASECAMP-1 (NCT04981119)
* Preconditioning lymphodepletion (PCLD) regimen
* A2B395 Tmod CAR T cells at the assigned dose

DETAILED DESCRIPTION:
This is a seamless phase 1/2, multi-center, open-label study that enrolls adults with recurrent unresectable, locally advanced, or metastatic (considered non-curative) CRC, NSCLC, HNSCC, TNBC, RCC, or other solid tumors with EGFR expression. Subjects must be germline HLA-A*02 heterozygous, with tumors that express EGFR and have lost HLA-A*02 expression. The purpose of Phase 1 of this study is to determine the safety and the optimal dose of A2B395 (after PCLD) in participants with solid tumor disease. The purpose of Phase 2 of this study is to determine the further safety and efficacy (how well it treats the solid tumor disease) of A2B395.

The treatment available for these cancers and other solid tumors can be toxic, debilitating, and fatal. In the recurrent unresectable, locally advanced, or metastatic setting, the intent of standard of care treatment is typically palliative rather than curative, and has not changed significantly in several decades. A2 Bio hypothesizes that A2B395 Tmod CAR T-cell therapy will enable the killing of tumor target cells (those cells that express EGFR and have loss of heterozygosity [LOH] for the HLA-A*02 protein). Additionally, normal healthy cells that maintain HLA-A*02 expression and co-express EGFR (eg, skin tissue) will not be targeted due to the blocker portion of the Tmod CAR T cell that acts as a self-regulated safety switch that protects normal tissue from damage. Furthermore, the blocker portion of the Tmod CAR T cell will act as a safety switch to protect normal tissue from graft versus host disease (GvHD) that could be caused by an allogeneic CAR T cell. A2 Bio intends this to provide a wider therapeutic safety window compared to previous solid tumor targeting therapies. This hypothesis will be explored in the study.

Participants for this study must enroll and have confirmation of LOH in the pre-screening BASECAMP-1 study (NCT04981119). Upon disease progression the participant may screen for this study (DENALI-1). There is no time requirement between the studies, and patients may go directly from BASECAMP-1 to DENALI-1 based on their own disease course.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Appropriately enrolled in the BASECAMP-1 A2 Biotherapeutics, Inc. study, with tissue demonstrating LOH of HLA-A*02 by NGS (whenever possible from the primary site).
2. Histologically confirmed recurrent unresectable, locally advanced, or metastatic CRC, NSCLC, HNSCC, TNBC, RCC, or other solid tumors with EGFR expression. Measurable disease is required with lesions of ≥1.0 cm by CT.
3. Received previous required therapy for the appropriate solid tumor disease as described in the protocol
4. Has adequate organ function as described in the protocol
5. ECOG performance status of 0 to 1
6. Life expectancy of ≥3 months
7. Willing to comply with study schedule of assessments including long-term safety follow-up

Key Exclusion Criteria:

1. Has disease that is suitable for local therapy or able to receive standard of care therapy that is therapeutic and not palliative
2. Prior allogeneic stem cell transplant
3. Prior solid organ transplant
4. Cancer therapy within 3 weeks or 3 half lives of A2B395 infusion
5. Radiotherapy within 28 days of A2B395 infusion
6. Unstable angina, arrhythmia, myocardial infarction, or any other significant cardiac disease within the last 6 months
7. Any new symptomatic pulmonary embolism (PE) or a deep vein thrombosis (DVT) within 3 months of enrollment. Therapeutic dosing of anticoagulants is allowed for history of PE or DVT if greater than 3 months from time of enrollment, and adequately treated
8. History of interstitial lung disease including drug-induced interstitial lung disease and radiation pneumonitis that requires treatment with prolonged steroids or other immune suppressive agents within 1 year
9. Requires supplemental home oxygen
10. Females of childbearing potential who are pregnant or breastfeeding
11. Subjects, both male and female, of childbearing potential who are not willing to practice birth control from the time of consent through 6 months post infusion of A2B395

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Rate of adverse events and dose limiting toxicities (DLTs) by dose level | From the time of Informed consent until 24 months (2 years) post A2B395 infusion
  Adverse events and toxicity will be evaluated according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (or current version). Cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), and graft versus host disease (GvHD) events will be graded according to the criteria described in the current protocol.
Phase 1: Recommended phase 2 dose (RP2D) | 28 days post A2B395 infusion
  The RP2D will be identified utilizing a BOIN study design in addition to considering safety and biomarker analysis.
Phase 2: The overall response rate (ORR) for patients | 24 months post A2B395 infusion
  The ORR will be evaluated per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and assessed by independent central review.

SECONDARY OUTCOMES:
Persistence of A2B395 | up to 24 months post A2B395 infusion
  Number of A2B395 Tmod CAR T cells present in participants treated with A2B395 as assessed by polymerase chain reaction (PCR) (or similar method) on participant blood samples
Cytokine analysis | up to 24 months post A2B395 infusion
  Cytokine levels such as interferon-gamma (IFN-γ) in participants treated with A2B395 assessed by cytokine analysis on participant blood samples
Cytokine analysis | up to 24 months post A2B395 infusion
  Cytokine levels such as interleukin-6 (IL-6) in participants treated with A2B395 assessed by cytokine analysis on participant blood samples

CONTACTS AND LOCATIONS:
Overall Officials: John Welch, MD, PhD, Study Director — A2 Biotherapeutics
Locations (10):
- United States (10):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Fred Hutch Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared within 1 year of study completion.
Supporting Information: CSR
Time Frame: Data will be available within 1 year of the completion of the study, the length of time of availability is to be determined.

REFERENCES:
- [Background] DiAndreth B, Hamburger AE, Xu H, Kamb A. The Tmod cellular logic gate as a solution for tumor-selective immunotherapy. Clin Immunol. 2022 Aug;241:109030. doi: 10.1016/j.clim.2022.109030. Epub 2022 May 11. PMID 35561999
- [Background] Oh J, Kirsh C, Hsin JP, Radecki KC, Zampieri A, Manry D, Ando Y, Miller S, Chan J, McLeod E, Cunningham KM, Wong LM, Xu H, Kamb A. NOT gated T cells that selectively target EGFR and other widely expressed tumor antigens. iScience. 2024 May 7;27(6):109913. doi: 10.1016/j.isci.2024.109913. eCollection 2024 Jun 21. PMID 38799557
- [Background] Beroukhim R, Mermel CH, Porter D, Wei G, Raychaudhuri S, Donovan J, Barretina J, Boehm JS, Dobson J, Urashima M, Mc Henry KT, Pinchback RM, Ligon AH, Cho YJ, Haery L, Greulich H, Reich M, Winckler W, Lawrence MS, Weir BA, Tanaka KE, Chiang DY, Bass AJ, Loo A, Hoffman C, Prensner J, Liefeld T, Gao Q, Yecies D, Signoretti S, Maher E, Kaye FJ, Sasaki H, Tepper JE, Fletcher JA, Tabernero J, Baselga J, Tsao MS, Demichelis F, Rubin MA, Janne PA, Daly MJ, Nucera C, Levine RL, Ebert BL, Gabriel S, Rustgi AK, Antonescu CR, Ladanyi M, Letai A, Garraway LA, Loda M, Beer DG, True LD, Okamoto A, Pomeroy SL, Singer S, Golub TR, Lander ES, Getz G, Sellers WR, Meyerson M. The landscape of somatic copy-number alteration across human cancers. Nature. 2010 Feb 18;463(7283):899-905. doi: 10.1038/nature08822. PMID 20164920
- [Background] Hwang MS, Mog BJ, Douglass J, Pearlman AH, Hsiue EH, Paul S, DiNapoli SR, Konig MF, Pardoll DM, Gabelli SB, Bettegowda C, Papadopoulos N, Vogelstein B, Zhou S, Kinzler KW. Targeting loss of heterozygosity for cancer-specific immunotherapy. Proc Natl Acad Sci U S A. 2021 Mar 23;118(12):e2022410118. doi: 10.1073/pnas.2022410118. PMID 33731480
- [Background] Hamburger AE, DiAndreth B, Cui J, Daris ME, Munguia ML, Deshmukh K, Mock JY, Asuelime GE, Lim ED, Kreke MR, Tokatlian T, Kamb A. Engineered T cells directed at tumors with defined allelic loss. Mol Immunol. 2020 Dec;128:298-310. doi: 10.1016/j.molimm.2020.09.012. Epub 2020 Oct 1. PMID 33012527
- See also: A2 Biotherapeutics Inc. — http://www.a2bio.com